CLINICAL TRIAL: NCT06841042
Title: A Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of SCTB35 in Patients with Systemic Lupus Erythematosus
Brief Title: A Study of SCTB35 in Patients with Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCTB35-X201
Record Dates: First submitted 2025-02-11; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: System Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: SCTB35 (Experimental): SCTB35 will be administered every 21 days per treatment cycle.
  Interventions: Biological: SCTB35 injection

INTERVENTIONS:
Biological: SCTB35 injection — SCTB35 will be subcutaneously administered at a dose as specified in the respective dose-escalation cohorts. Then, the RP2D and other appropriate doses of SCTB35 will be applied for the dose-expansion cohorts.

SUMMARY:
This study is a multicenter Phase Ib/II clinical trial aimed at evaluating the safety, tolerability and efficacy of SCTB35 in patients with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This study contains the dose-escalation and dose-expansion parts. The escalation cohorts will be enrolled to explore the maximum tolerated dose and recommended phase II dose (RP2D). A Safety Review Committee (SRC) will review the accumulated safety data and other available data, and make a recommendation to each dose level of SCTB35 in the escalation cohorts. The expansion cohorts will be initiated after the RP2D is confirmed, and to further compare the preliminary efficacy and safety of SCTB35 at appropriate dose levels recommended by SRC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years；
2. Diagnosed with SLE for ≥12 weeks prior to screening (2019-ACR/EULAR criteria);
3. SLEDAI-2K ≥ 8 at screening, or ≥6 if there is hypocomplementemia or elevated anti-dsDNA antibody levels;
4. Positive for ANA (1:80) or positive for anti-dsDNA and/or anti-Sm antibodies within the last 12 months or at screening;
5. Currently receiving ≥1 stable dose of standard treatment: oral corticosteroids, antimalarials, or conventional immunosuppressive drugs

   1. Stable corticosteroid dose for ≥4 weeks prior to baseline;
   2. Stable dose of antimalarial drugs for ≥4 weeks prior to baseline;
   3. Stable dose of immunosuppressive agents for ≥4 weeks prior to baseline;
6. All male participants or females of reproductive potential must agree to use reliable contraception with their partner from signing the ICF through 6 months after the last dose of the study drug;
7. Understanding of the study procedures and voluntary signing of the informed consent form.

Exclusion Criteria:

1. Severe active or unstable lupus-related neuropsychiatric disorders;
2. Other autoimmune diseases that may interfere with efficacy evaluation;
3. Catastrophic antiphospholipid syndrome;
4. Received treatments that may affect the drug's effect:
5. Received live vaccines or attenuated vaccines within 28 days prior to baseline or screening;
6. Clinically significant bleeding risk;
7. Abnormal laboratory results:

   1. AST or ALT >2.5 x ULN;
   2. Total bilirubin >1.5 x ULN;
   3. ANC <1.5x10⁹/L;
   4. Platelets <75x10⁹/L;
   5. Hemoglobin <100g/L;
8. eGFR <30 mL/min/1.73 m²;
9. Positive serum HCG;
10. Received any investigational treatment within 30 days prior to baseline or within 5 half-lives of the investigational drug (whichever is longer);
11. Participants with recurrent, chronic, or other active infections as assessed by the investigator;
12. Severe or uncontrolled disease, which would prevent participation in the study;
13. Positive viral serology tests, including HIV, HCV, and HBV;
14. Tuberculosis screening: Known active tuberculosis or latent tuberculosis infection (LTBI);
15. Any type of active infection except nail bed fungal infections;
16. Severe infections;
17. History of progressive multifocal leukoencephalopathy (PML);
18. Diagnosed with type 1 or type 2 diabetes with poor control;
19. Uncontrolled hypertension (systolic >140 mmHg or diastolic >90 mmHg);
20. History of malignancy within 5 years prior to baseline;
21. Alcohol abuse or drug misuse within 12 months prior to screening;
22. Intolerance to the study drug or contraindications, including a history of severe allergic reactions to monoclonal antibodies or any component of SCTB35 injection;
23. Required hospitalization for major surgery within 4 weeks prior to screening or within 12 weeks post-study drug administration;
24. Participants with mental disorders or poor compliance;
25. Severe lupus nephritis;
26. History of solid organ or hematopoietic stem cell/bone marrow transplant, or expected to undergo transplant surgery during the study;
27. Pregnant or breastfeeding;
28. Any other condition that the investigator deems unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Dose-escalation part： Incidence rate of adverse event (AE) | From first dose to the 24 weeks
  To evaluate the incidence rates of treatment emergent adverse event (TEAE), treatment-related TEAE (TRAE), serious adverse event (SAE), adverse event with special interest (AESI)
Dose-expansion part：SRI-4 | Up to Week 24
  Percentage of subjects who achieved an SRI-4 response at 24 weeks；

SECONDARY OUTCOMES:
Dose-escalation part： SLEDAI-2K | Up to week 12, 24
  Percentage of subjects with a reduction of ≥4 points in SLEDAI-2K at 12 and 24 weeks.
Dose-escalation part： physician global assessment (PGA) | Up to week 12, 24
  Percentage of subjects with no worsening in PGA, where worsening is defined as a ≥0.3 point increase in PGA at 12 and 24 weeks.
Dose-escalation part：Immunogenicity； | From baseline to Week 24
  Serum anti-SCTB35 antibody and anti-SCTB35 antibody levels before and after administration
Dose-expansion part：SLEDAI-2K | Up to week 12, 24
  Percentage of subjects with a reduction of ≥4 points in SLEDAI-2K at 12 and 24 weeks.
Dose-expansion part： BILAG | Up to week 12, 24
  Percentage of subjects with no new BILAG A or ≤1 new BILAG B at 12 and 24 weeks.
Dose-expansion part： PGA | Up to week 12, 24
  Percentage of subjects with no worsening in PGA at 12 and 24 weeks.
Dose-expansion part： SFI | Up to week 52
  Time to first disease relapse

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Jilin Provincial People's Hospital, Changchun
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First People's Hospital of Jiujiang City, Jiujiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming
  - Linfen Central Hospital, Linfen
  - Mianyang Central Hospital, Mianyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Pingxiang People's Hospital, Pingxiang
  - Shanxi Bethune Hospital, Taiyuan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xinxiang Central Hospital, Xinxiang

IPD SHARING:
Plan to Share IPD: Undecided